CLINICAL TRIAL: NCT03788382
Title: Failure to Adjuvant Therapy After Pancreatic Resection for Pancreatic Cancer: a Real Life Scenario
Brief Title: Failure to Adjuvant Therapy After Pancreatic Resection for Pancreatic Cancer
Acronym: FOUNTAIN
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Salvatore Paiella, MD, Salvatore Paiella, MD, Università di Verona, Universita di Verona
Other Study IDs: FOUNTAIN
Record Dates: First submitted 2018-12-21; First posted 2018-12-27 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Malignant Neoplasm Primary
Keywords: Failure Adjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the rate of patients submitted to pancreatic resection for pancreatic cancer, who fail to access to adjuvant therapy or do not complete adjuvant therapy. The purpose is to give an overview concerning the most frequent conditions and/or reasons associated with failure or omission of adjuvant therapy.

DETAILED DESCRIPTION:
This prospective observational study will evaluate all patients submitted to pancreatic resection for pancreatic cancer.

The rate of omission to adjuvant therapy and rate of failure of completion of adjuvant therapy will be evaluated as primary outcomes. As secondary outcomes, survival analyses will be performed to investigate whether these factors influence prognosis, that will be evaluated through a disease free survival analysis at 18-months. Epidemiological and perioperative data will be analyzed to identify conditions associated with the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of pancreatic cancer

Exclusion Criteria:

* Non exocrine pancreatic tumors
* Periampullary malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to Pancreatic Resection for Pancreatic Cancer
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Rate of patients who fail to receive adjuvant therapy and reasons for that | 6 months
  The amount of patients who will not receive adjuvant therapy after pancreatic resection for malignancy (when do indication exists) will be recorded
Rate of patients who fail to complete adjuvant therapy and reasons for that | 9 months
  The amount of patients who will not complete adjuvant therapy after pancreatic resection for malignancy will be recorded

SECONDARY OUTCOMES:
Disease free survival of patients enrolled | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona Hospital, Verona, Italy

REFERENCES:
- [Derived] Paiella S, Malleo G, Lionetto G, Cattelani A, Casciani F, Secchettin E, De Pastena M, Bassi C, Salvia R. Adjuvant Therapy After Upfront Resection of Resectable Pancreatic Cancer: Patterns of Omission and Use-A Prospective Real-Life Study. Ann Surg Oncol. 2024 May;31(5):2892-2901. doi: 10.1245/s10434-024-14951-4. Epub 2024 Jan 29. PMID 38286884